CLINICAL TRIAL: NCT02490072
Title: Echocardiographic Evaluation of the Effects of Dexmedetomidine in Diastolic Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double
Other Study IDs: 4-2015-0284
Record Dates: First submitted 2015-06-15; First posted 2015-07-03 (Estimated); Last update posted 2015-08-10 (Estimated); Status verified 2015-08

CONDITIONS: Under General Anesthesia
MeSH Terms: interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexmedetomidine group (Experimental)
  Interventions: Drug: Dexmedetomidine
- normal saline (Placebo Comparator)
  Interventions: Drug: normal saline(Saline 0.9%)

INTERVENTIONS:
Drug: Dexmedetomidine — Formula for administrated were randomized by computer-generated randomization. The patients and anesthesiologist, who administered and conducted all this trial, were blinded to the medication allocation. An anesthesiologist, who responsible for preparation of medication was the only person, recognized of the randomization code during trial. 10 minutes after anesthetic induction, dexmedetomidine group would start the loading of dexmedetomidine (1μg/kg) during 10 minutes followed infusion of dexmedetomidine(0.5 μg/kg/min). Bispectral index was monitored continuously targeting 40±5. Target concentration of remifentanil and fresofol were controlled stepwise in accordance with BIS. Using the transesophageal echocardiography, we will evaluate the changes of cardiac function including Tei index and cardiac output.
  Arms: Dexmedetomidine group
Drug: normal saline(Saline 0.9%)
  Arms: normal saline

SUMMARY:
Dexmedetomidine is a selective α2 adrenergic agonist that can be considered a primary anesthetic, an adjuvant to propofol or inhalational anesthetics. Dexmedetomidine mediate its cardiovascular effect through activation of receptors in central and peripheral nervous system. The classic cardiovascular response of dexmedetomidine is the biphasic with initial shorten-increase in blood pressure followed by long-lasting decrease in BP and HR. There were several reports about these hemodynamic changs of dexmedetomidine, but not the evaluation of direct cardiac function of patients who was preexisted diastolic dysfunction. The purpose of this study is to evaluate the effects of dexmedetomidine as an anesthetic adjuvant in diastolic dysfunction by using the echocardiography.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria included patients who estimated lateral e' velocity <10 cm/s or septal e' velocity <8 cm/s from the mitral annuli and averaged E/e' ≧ 9 in preoperative echocardiographic evaluation. For patients of old age (> 60 yr) who did not undergo preoperative echocardiographic evaluation, written consent was obtained and TTE was performed to evaluate presence of diastolic dysfunction; patients with diastolic dysfunction, as previous defined, were included and those without were excluded

1. Above 40 years of age.
2. American Society of Anesthesiologists (ASA) Physical Status II, III.
3. Preserved systolic function (Ejection fraction > 50%)

Exclusion Criteria:

The exclusion criteria included patients who estimated lateral e' velocity >10 cm/s or septal e' velocity >8 cm/s from the mitral annuli, and averaged E/e' ≦ 8 in preoperative echocardiographic evaluation.

1. severe functional liver or kidney disease
2. diagnosed HF (LV ejection fraction <50% , or wall motion abnormality)
3. arrhythmia or received treatment with antiarrythmic drug .
4. severe bradycardia(HR < 45 bpm) and AV block 6. pathologic esophageal lesion (esophageal stricture or varix ) 7. pregnancy 8. severe chronic obstructive lung disease.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-07; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
biventricular diastolic function | Change from baseline 10 min after induction (T1), 20 min after Dex loading (T2), 40 min after Dex loading (T3), 60 min after Dex loading(T4)
  E/e'estimated by using tissue Doppler index

SECONDARY OUTCOMES:
Tei-index (myocardial performance index) | Change from baseline 10 min after induction(T1), 20 min after Dex loading (T2), 40 min after Dex loading (T3), 60 min after Dex loading(T4)
  tissue Doppler image-derived myocardial performance

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institue, Yonsei Universiy College of Medicine, Seoul, Seoul, South Korea